CLINICAL TRIAL: NCT06673888
Title: Clinical Assessment of an Alkasite-Based Resin Composite Restorative Material Versus Resin Modified Glass Ionomer-Based Restorative Material in Class V Cavities: One Year Randomized Clinical Trial
Brief Title: Assessment of Alkasite Restorative Material Versus Resin Modified Glass Ionomer in Class V Cavities: a Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Mokhtar Anwar Ismail, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cention Forte Protocol
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Class V Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alkasite-Based Resin Composite Restorative Material (Bioactive Material) (Experimental): Alkasite material releases hydroxyl ions, calcium, fluoride, and phosphate ions which explains its caries-prevention mechanisms. Many researches indicate that this alkasite material neutralizes acids and prevents enamel and dentin demineralization when exposed to lactic acid for an extended length of time together with the added advantageous of maximum properties and esthetics of resin composite
  Interventions: Other: alkasite based restorative material
- Resin Modified Glass Ionomer Restorative Material (Active Comparator): Resin-modified glass-ionomers have mainly the same clinical applications as conventional glass-ionomers. Their biocompatibility and ability to release fluoride are two of their advantages. In addition, it has advantages over traditional glass ionomer in terms of stronger features, better aesthetics, earlier finishing, and longer working time. They are considered the gold standard in restoring cervical carious lesions of anterior teeth over GI due to their added benefit of higher esthetics.
  Interventions: Other: Resin modified glass ionomer

INTERVENTIONS:
Other: Resin modified glass ionomer — Resin modified glass ionomer (RMGI) is utilized for a variety of purposes, as luting agents, liners/bases, and restorative materials. The RMGI is more aesthetically pleasing than the conventional glass ionomer while maintaining the clinical benefits of the former, such as the release of fluoride, recharging capabilities, prevention of decalcification of hard tooth tissue, inhibition of bacterial acid metabolism, and ease of clinical operation.
  Arms: Resin Modified Glass Ionomer Restorative Material
Other: alkasite based restorative material — Cention forte is bioactive restorative material which has the ability to remineralize hard dental tissues through calcium and fluoride release and can also neutralize bacterial acids through hydroxide ions release.
  Arms: Alkasite-Based Resin Composite Restorative Material (Bioactive Material)

SUMMARY:
This study will be conducted to evaluate the clinical assessment of an alkasite based resin composite restorative material compared to resin modified glass ionomer based restorative material in class V cavities of anterior teeth over 12 months follow up using modified USPHS criteria.

In patients with anterior cervical (class V) carious lesions, will the novel alkasite-based restorative material show similar clinical assessment as resin modified glass ionomer over a one year follow up period?

DETAILED DESCRIPTION:
Dental caries is a common chronic infectious illness caused by cariogenic bacteria that metabolize sugars to generate acid, which gradually demineralizes tooth structure. Dental caries is a major healthcare problem as it is the most prevalent disease worldwide. Low socioeconomic level groups are more likely to be affected by the disease and during the past thirty years, its prevalence has not considerably decreased despite being completely preventable.

Non-invasive methods (such as sealing, biofilm removal, and remineralization) should be used to treat existing early caries rather than removing the dental tissue. Cavitated lesions should be arrested or managed using a minimally invasive method, such as conservative cavity designs, and repairing defective restoration rather than replacing it.

Ion-releasing restorations are recognized for their biocompatibility with surrounding tissues and their fluoride-releasing capabilities, which are thought to help prevent caries by creating an oral environment that prevents the demineralization of surrounding hard tooth tissue.

Resin modified glass ionomer (RMGI) is utilized for a variety of purposes, as luting agents, liners/bases, and restorative materials. The RMGI is more aesthetically pleasing than the conventional glass ionomer while maintaining the clinical benefits of the former, such as the release of fluoride, recharging capabilities, prevention of decalcification of hard tooth tissue, inhibition of bacterial acid metabolism, and ease of clinical operation.

A novel family of bioactive "alkasite" restorative materials, essentially a subgroup of composite resin, represents a new era of restorative dentistry. This material is available in a capsulated form using a unique adhesive system. An alkaline filler that has the ability to release ions that neutralize acids is used in this novel material. It is stated that this substance can neutralize bacterial acids by releasing hydroxide ions and remineralize hard dental tissues by releasing calcium and fluoride. The material's release of ions may be crucial in neutralizing the effects of cariogenic bacteria, thus guarding against tooth caries.

The author conducted a study to evaluate the performance of two different restorative materials in patients with class V carious lesion in upper anterior teeth where the esthetic appearances is highly recommended.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (30-40Ys) with class V cavities (ICDAS 4 or 5) in upper anterior teeth.

  * Males or females.
  * Have sufficient cognitive ability to understand consent procedures.
  * Co-operative patients approving to participate in the trial.
  * Anterior tooth cervical carious lesion with ICDAS score 4 or 5.
  * Vital upper anterior teeth with no signs or symptoms of irreversible pulpitis.
  * Mobility grade: no clinical mobility.
  * Teeth with healthy periodontium.

Exclusion Criteria:

* • Disabilities.

  * Systemic diseases or severe medically compromised.
  * Lack of compliance.
  * Evidence of severe bruxism, clenching or temporomandibular joint disorders.
  * Cognitive impairment
  * Periapical pathosis or signs of pulpal pathology.
  * Non-vital tooth.
  * Signs of pathological wear.
  * Endodontically treated tooth.
  * Severe periodontal affection or tooth indicated for extraction.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical assessment | 12 months change from base line to six and 12 months.
  clinical assessment of retention, color match , Marginal Adaptation, marginal discoloration , Anatomical form ,Surface texture, secondary caries and postoperative hypersensitivity , All these outcomes are measured using modified USPH criteria for clinical evaluation of restoration failure where they are given scores Alpha is excellent , Bravo is acceptable ,Charlie is not accepted.

IPD SHARING:
Plan to Share IPD: No